CLINICAL TRIAL: NCT01962298
Title: Sugammadex and the Diaphragm: Recovery of Diaphragmatic Function and Neuromuscular Blockade. A Double-blind Randomized Controlled Trial
Brief Title: Recovery of Diaphragmatic Function After Neuromuscular Blockade and Sugammadex
Acronym: SUDIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Tom Schepens, MD, Tom Schepens, MD, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC 13/5/60; 2013-001926-25 (EudraCT Number); B300201316844 (Registry Identifier: Belgisch Registratienummer)
Record Dates: First submitted 2013-10-09; First posted 2013-10-14 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-03

CONDITIONS: Diaphragmatic Dysfunction; Muscle Weakness; Muscle Fatigue
MeSH Terms: conditions — Muscle Weakness | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Single rocuronium dose - placebo (Placebo Comparator): The patients will receive a single rocuronium dose, and no reversal agent.
  Interventions: Drug: placebo; Drug: Single rocuronium dose
- Single rocuronium dose - sugammadex (Active Comparator): The patients will receive a single rocuronium dose and sugammadex 2mg/kg as a reversal agent
  Interventions: Drug: sugammadex 2mg/kg; Drug: Single rocuronium dose
- Repeated rocuronium dose - neostigmine (Active Comparator): The patients will receive multiple rocuronium doses and neostigmine 70 mcg/kg as a reversal agent
  Interventions: Drug: neostigmine; Drug: Repeated rocuronium dose
- Repeated rocuronium dose - sugammadex (Active Comparator): The patients will receive multiple rocuronium doses and neostigmine 2mg/kg as a reversal agent
  Interventions: Drug: sugammadex 2mg/kg; Drug: Repeated rocuronium dose
- Continuous rocuronium dose (Active Comparator): The participants will receive a continuous rocuronium infusion and sugammadex 4 mg/kg as a reversal agent
  Interventions: Drug: sugammadex 4mg/kg; Drug: Continuous rocuronium infusion

INTERVENTIONS:
Drug: sugammadex 2mg/kg
  Arms: Repeated rocuronium dose - sugammadex; Single rocuronium dose - sugammadex
Drug: neostigmine
  Arms: Repeated rocuronium dose - neostigmine
Drug: sugammadex 4mg/kg
  Arms: Continuous rocuronium dose
Drug: placebo
  Arms: Single rocuronium dose - placebo
Drug: Single rocuronium dose
  Arms: Single rocuronium dose - placebo; Single rocuronium dose - sugammadex
Drug: Repeated rocuronium dose
  Arms: Repeated rocuronium dose - neostigmine; Repeated rocuronium dose - sugammadex
Drug: Continuous rocuronium infusion
  Arms: Continuous rocuronium dose

SUMMARY:
The effect of neuromuscular blocking agents (NMBA, e.g. rocuronium) on respiratory muscle activity is well known. However, since the availability of sugammadex, to our knowledge, no study has been conducted to evaluate the effect of this novel product on these muscles.

Our hypothesis is that by applying a different strategy in the use of neuromuscular blocking agents and their reversal agents we might see a different activity of the respiratory muscles.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must have the mental capacity to decide whether he/she takes part in the trial or not. Each participant must voluntarily give his/her written informed consent. In case a participant is physically unable to give a written informed consent, a legal representative is to perform this.
* Each participant must be at least eighteen years of age. Participants can be of either sex and of any ethnical background.
* Each participant must meet the American Society of Anesthesiologists class II, II or III criteria.
* Each participant must be scheduled for intracranial surgery. During general anesthesia rocuronium must be used as a neuromuscular blocking agent.
* Each participant must be a suitable candidate for the rapid reversal of the neuromuscular blockade.
* Each female participant of sexually active age and of childbearing potential must agree to the use of a medically accepted method of contraception through seven days after the day of surgery. Postmenopausal (defined as at least twelve consecutive months without spontaneous menstrual period) women are not obliged to use contraceptives.

Exclusion Criteria:

* The participant is known or suspected to have a neuromuscular disorder.
* The participant is known or suspected to have an allergic reaction to sugammadex, rocuronium, anesthetic or narcotic medications, or any drugs used during general anesthesia.
* The participant is known or suspected to have an anatomical malformation impeding a proper intubation.
* The participant is known or suspected to have a history of malignant hyperthermia.
* The participant is pregnant (or intends to become pregnant within the presurgical period) or lactating.
* The participant is known to have a renal insufficiency (defined as a serum creatinine concentration of two times the upper limit, or a glomerular filtration rate of less than 60 ml/min).
* The participant is known or suspected to have a chronic obstructive pulmonary disease GOLD classification 2 or higher or has any respiratory disease that impairs his respiratory function to a NYHA III level or worse.
* The participant is known to have an infection of the upper or lower airways, as diagnosed by clinical or laboratory findings.
* The participant is known or suspected to have congestive heart failure.
* The participant is obese, as defined by a body mass index of 30 kg/m2 or more.
* The participant is known or suspected to have a major hepatic dysfunction.
* The participant has received or is scheduled to receive toremifene and/or an intravenous administration of fusidic acid within a time span of twenty-four hours before and twenty-four hours after the surgery.
* The participant is known or suspected to have any condition contraindicating the administration of sugammadex, neostigmine, glycopyrrolate or placebo.
* The participant is known or suspected to be directly involved in this study and/or is employed by or is a family member of any person employed by the investigator, at the investigational site, or by the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerpen, Belgium

REFERENCES:
- [Background] Dres M, Schmidt M, Ferre A, Mayaux J, Similowski T, Demoule A. Diaphragm electromyographic activity as a predictor of weaning failure. Intensive Care Med. 2012 Dec;38(12):2017-25. doi: 10.1007/s00134-012-2700-3. Epub 2012 Sep 26. PMID 23011532
- [Derived] Schepens T, Janssens K, Maes S, Wildemeersch D, Vellinga J, Jorens PG, Saldien V. Respiratory muscle activity after spontaneous, neostigmine- or sugammadex-enhanced recovery of neuromuscular blockade: a double blind prospective randomized controlled trial. BMC Anesthesiol. 2019 Oct 19;19(1):187. doi: 10.1186/s12871-019-0863-y. PMID 31629404

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for inclusion and approached the night prior to their elective surgery
Groups:
- Single Rocuronium Dose - Placebo: The patients will receive a single rocuronium dose, and no reversal agent.
  placebo
  Single rocuronium dose
- Single Rocuronium Dose - Sugammadex: The patients will receive a single rocuronium dose and sugammadex 2mg/kg as a reversal agent
  sugammadex 2mg/kg
  Single rocuronium dose
- Repeated Rocuronium Dose - Neostigmine: The patients will receive multiple rocuronium doses and neostigmine 50 mcg/kg as a reversal agent
  neostigmine
  Repeated rocuronium dose
- Repeated Rocuronium Dose - Sugammadex: The patients will receive multiple rocuronium doses and neostigmine 2mg/kg as a reversal agent
  sugammadex 2mg/kg
  Repeated rocuronium dose
- Continuous Rocuronium Dose: The participants will receive a continuous rocuronium infusion and sugammadex 4 mg/kg as a reversal agent
  sugammadex 4mg/kg
  Continuous rocuronium infusion
Period: Overall Study
Arm/Group | Single Rocuronium Dose - Placebo | Single Rocuronium Dose - Sugammadex | Repeated Rocuronium Dose - Neostigmine | Repeated Rocuronium Dose - Sugammadex | Continuous Rocuronium Dose
Started | 15 | 15 | 15 | 15 | 15
Received Intervention | 14 (1 subject did not receive the planned intervention and received a different one for clinical reasons) | 15 | 15 | 15 | 15
Completed | 12 | 11 | 10 | 13 | 9
Not Completed | 3 | 4 | 5 | 2 | 6
Not completed — Protocol Violation | 1 | 0 | 1 | 1 | 0
Not completed — Data quality insufficient | 2 | 0 | 3 | 1 | 4
Not completed — Insufficient data | 0 | 2 | 1 | 0 | 1
Not completed — Incorrect data recorded | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Rocuronium Dose - Placebo | Single Rocuronium Dose - Sugammadex | Repeated Rocuronium Dose - Neostigmine | Repeated Rocuronium Dose - Sugammadex | Continuous Rocuronium Dose | Total
Number analyzed (Participants) | 12 | 11 | 10 | 13 | 9 | 55
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [42 to 63] | 51 [41 to 65] | 56 [49 to 59] | 54 [30 to 68] | 55 [41 to 63] | 55 [44 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 6 | 7 | 6 | 33
  Male | 6 | 3 | 4 | 6 | 3 | 22
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m2] | 26 [23 to 30] | 27 [24 to 28] | 25 [21 to 28] | 26 [24 to 28] | 24 [21 to 27] | 26 [22 to 28]

OUTCOME MEASURES:

1. Primary Outcome: Electric Activity of the Diaphragm (Microvolts)
Time Frame: From the start of spontaneous breathing till extubation, limited to maximum ten minutes after the onset of spontaneous breathing
Measure: Median (Inter-Quartile Range); unit: microvolt
Arm/Group | Single Rocuronium Dose - Placebo | Single Rocuronium Dose - Sugammadex | Repeated Rocuronium Dose - Neostigmine | Repeated Rocuronium Dose - Sugammadex | Continuous Rocuronium Dose
Number analyzed (Participants) | 12 | 11 | 10 | 13 | 9
microvolt | 3.7 [1.7 to 7.7] | 4.5 [2.1 to 8.0] | 3.2 [0.9 to 7.3] | 2.9 [1.3 to 5.3] | 4.4 [1.9 to 7.5]

2. Secondary Outcome: Electric Activity of the Intercostal Muscles
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: microvolt
Arm/Group | Single Rocuronium Dose - Placebo | Single Rocuronium Dose - Sugammadex | Repeated Rocuronium Dose - Neostigmine | Repeated Rocuronium Dose - Sugammadex | Continuous Rocuronium Dose
Number analyzed (Participants) | 12 | 11 | 10 | 13 | 9
microvolt | 2.4 [1.4 to 4.5] | 2.2 [1.2 to 4.7] | 1.5 [1.1 to 2.5] | 2.2 [1.3 to 4.5] | 1.8 [1.1 to 3.7]

3. Other Pre Specified Outcome: Centroid Frequency of the EMG, as Trend Variability (Change in %) From First to Last Recording
Time Frame: From the start of spontaneous breathing till extubation, limited to maximum one hour after the onset of spontaneous breathing
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Single Rocuronium Dose - Placebo | Single Rocuronium Dose - Sugammadex | Repeated Rocuronium Dose - Neostigmine | Repeated Rocuronium Dose - Sugammadex | Continuous Rocuronium Dose
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes